CLINICAL TRIAL: NCT02898857
Title: CHEMO RESISTANCE TO PLATINUM COMPOUNDS AND NOTCH PATHWAYS IN PATIENTS RECEIVING NEOADJUVANT CHEMOTHRERAPY FOR LOCALLY ADVANCED ADENOCARCINOMA OF THE LUNG.
Brief Title: Chemoresistance and Involvement of the NOTCH Pathway in Patients With Lung Adenocarcinoma
Acronym: NOTCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut de Recherche en Cancérologie de Montpellier (IRCM) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 9758
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Biopsy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- down-staging of a KRAS: Six with demonstrated down-staging of a KRAS mutant adenocarcinoma who underwent biopsie The biopsies of lung tumour samples will be analysed by immunochemistry (IHC), western blotting and qPolymerase Chain Reaction (PCR) approaches
  Interventions: Other: biopsies
- no down-staging of a KRAS: Six with demonstrated no down-staging (persistent tumour cell involving lymph nodes in surgically resected specimens) of a KRAS mutant adenocarcinoma who underwent biopsie The biopsies of lung tumour samples will be analysed by immunochemistry (IHC), western blotting and qPolymerase Chain Reaction (PCR) approaches
  Interventions: Other: biopsies
- non-staging and triple negative adenocarcinoma: Six with or without non-staging and triple negative adenocarcinoma who underwent biopsie The biopsies of lung tumour samples will be analysed by immunochemistry (IHC), western blotting and qPolymerase Chain Reaction (PCR) approaches
  Interventions: Other: biopsies

INTERVENTIONS:
Other: biopsies — The biopsies of lung tumour samples will be analysed by immunochemistry (IHC), western blotting and qPolymerase Chain Reaction (PCR) approaches in Six with demonstrated down-staging of a KRAS mutant adenocarcinoma, Six with demonstrated no down-staging (persistent tumour cell involving lymph nodes in surgically resected specimens) of a KRAS mutant adenocarcinoma and Six with or without non-staging and triple negative adenocarcinoma

SUMMARY:
Every year in France, 30.000 deaths are due to lung cancer and 39.500 new cases of this disease are diagnosed (INCa 2014). Patients suffering from locally advanced non-small-cell lung cancer (NSCLC), stage IIIa, usually undergo a multimodality treatment including chemotherapy with platinum compounds before surgery (called neoadjuvant chemotherapy or induction chemotherapy). The reason of this combined modality treatment is the really poor prognosis of patients presenting a disease already spread to lymph nodes (classified N2 when the lymph node under the carina is affected). Up till now, the five-year survival of patients who underwent surgical resection of N2 NSCLC does not exceed 15%

DETAILED DESCRIPTION:
Every year in France, 30.000 deaths are due to lung cancer and 39.500 new cases of this disease are diagnosed (INCa 2014). Patients suffering from locally advanced non-small-cell lung cancer (NSCLC), stage IIIa, usually undergo a multimodality treatment including chemotherapy with platinum compounds before surgery (called neoadjuvant chemotherapy or induction chemotherapy). The reason of this combined modality treatment is the really poor prognosis of patients presenting a disease already spread to lymph nodes (classified N2 when the lymph node under the carina is affected). Up till now, the five-year survival of patients who underwent surgical resection of N2 NSCLC does not exceed 15%.

NOTCH pathway seems to be implicated in the resistance of tumor to chemotherapy. It is known that NOTCH plays a role in the homeostasis of adult stem cells and of cancer stem cells, including intestine cancer and NSCLC. In breast cancer, it has been demonstrated that NOTCH 1 plays a role in the relapse and adding a treatment by an inhibitor of NOTCH decreases the recurrence rate. An activation of the NOTCH pathway was proven in human lung cancer cell lines (A549 and H460) treated with cisplatin. Furthermore, HES1 (Hairy enhance of split), a downstream gene resulting from NOTCH transcription, was upregulated in patient with relapse comparing resistant versus non-resistant adenocarcinoma NSCLC patients. It was proved, NOTCH pathway is associated with overall survival in NSCLC. Recently, it was showed that an inhibitor of NOTCH combined with chemotherapy strongly potentiates the anti-tumor effects of the systemic therapy. Therefore, one can hypothesize that platinum compound-induced NOTCH activation contributes to the resistance of NSCLC and beyond this point, to tumor progression.

ELIGIBILITY:
Inclusion Criteria:

patients of both sex, aged 75 years or younger, diagnostic specimen demonstrating an adenocarcinoma, KRAS mutation on exon 2 and codon 12 or codon 13 or triple negative, clinical pathological N2, having received a platinum-based regimen as first line therapy, at less three courses of chemotherapy must have been delivered, with only these molecules : cisplatin-vinorelbine, cisplatin-gemcitabine, cisplatin-docetaxel, cisplatin-paclitaxel, having been operated upon and having been surgically resected R0 or R1.

Exclusion Criteria:

patients having received more than one line of preoperative chemotherapy, having received concurrent chemo-radiotherapy as preoperative treatment, no available diagnostic specimen, patients who underwent R2 resection or no resection, patients affected by adenocarcinoma harbouring either EGFR mutation or EML4-ALK translocation, patients with pathological complete response (yT0yN0).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Six with demonstrated down-staging of a KRAS mutant adenocarcinoma
  * Six with demonstrated no down-staging (persistent tumour cell involving lymph nodes in surgically resected specimens) of a KRAS mutant adenocarcinoma
  * Six with or without non-staging and triple negative adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
analysed by immunochemistry (IHC) | 1 day
  The biopsies of lung tumour samples will be analysed by immunochemistry (IHC)

SECONDARY OUTCOMES:
western blotting (WB) | 1 day
  The biopsies of lung tumour samples will be analysed by western blotting (WB)
qPolymerase Chain Reaction (PCR) | 1 day
  The biopsies of lung tumour samples will be analysed by qPolymerase Chain Reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PUJOL, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- PUJOL, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided